CLINICAL TRIAL: NCT01382316
Title: Making Alcoholics Anonymous Easier: A Group TSF Approach
Brief Title: Making Alcoholics Anonymous Easier
Acronym: MAAEZ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcohol Research Group (Other)
Responsible Party: Lee Ann Kaskutas, Alcohol Research Group, Public Health Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AA014688 (NIH); NCT01244919 (obsolete NCT alias)
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Alcohol Dependence; Drug Dependence
Keywords: 12-step facilitation; Alcoholics Anonymous; Narcotics Anonymous; AA; Self-help
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Making Alcoholics Anonymous Easier (Experimental): Six session, group format intervention, consisting of introductory session, four core sessions (sponsorship, principles not personalities, spirituality, living sober), and return to introductory session as MAAEZ graduate
  Interventions: Behavioral: Making Alcoholics Anonymous Easier (MAAEZ)
- Usual care (Active Comparator): Usual group sessions on education about alcohol and drug problems
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Making Alcoholics Anonymous Easier (MAAEZ) — 6-week, 90-minute, manualized, 12-step facilitation intervention consisting of 6 weekly session. First session is introduction. Four following core sessions attended in any order: sponsorship, principles not personalities, spirituality, living Sober. Last session, return to intro session as graduate.
  Other Names: MAAEZ
  Arms: Making Alcoholics Anonymous Easier
Behavioral: Usual care — Group format, six weekly education sessions about alcohol and drugs
  Arms: Usual care

SUMMARY:
This study tests the effectiveness of Making Alcoholics Anonymous Easier (MAAEZ), a manual-guided intervention designed to help alcohol and drug dependent clients connect with individuals encountered in AA. An OFF/ON design was used (n=508). MAAEZ effectiveness was determined by comparing abstinence rates of participants recruited during ON (MAAEZ intervention) and OFF (usual care) conditions and by studying the effect of the number of MAAEZ sessions attended. Better outcomes were hypothesized for MAAEZ vs. usual care. At 12 months, more clients in the ON condition (vs. OFF) reported past 30-day abstinence from alcohol, drugs, and both alcohol and drugs. Abstinence increased for each additional MAAEZ session received. MAAEZ appeared especially effective for those with more prior AA exposure, severe psychiatric problems, and atheists/agnostics. Mechanisms of action for MAAEZ (mediators of the MAAEZ effect) include: doing service in AA/NA/CA; having a sponsor; having a social network supportive of abstinence; and comfort being in meetings. MAAEZ represents an evidence-based intervention that is easily implemented in existing treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* current alcohol or drug dependence diagnosis

Exclusion Criteria:

* incapacitating mental or physical health; under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2005-07; Primary Completion 2006-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Alcohol and drug abstinence | Past 30 days
  No alcohol and no drug consumed during the 30 days prior to 12-month follow-up interview

CONTACTS AND LOCATIONS:
Overall Officials: Lee A Kaskutas, Dr.P.H., Principal Investigator — Alcohol Research Group, Public Health Institute
Locations (1):
- Alcohol Research Group, Emeryville, California, United States

REFERENCES:
- [Background] Kaskutas LA, Subbaraman MS, Witbrodt J, Zemore SE. Effectiveness of Making Alcoholics Anonymous Easier: a group format 12-step facilitation approach. J Subst Abuse Treat. 2009 Oct;37(3):228-39. doi: 10.1016/j.jsat.2009.01.004. Epub 2009 Apr 1. PMID 19339148
- [Background] Subbaraman MS, Kaskutas LA, Zemore S. Sponsorship and service as mediators of the effects of Making Alcoholics Anonymous Easier (MAAEZ), a 12-step facilitation intervention. Drug Alcohol Depend. 2011 Jul 1;116(1-3):117-24. doi: 10.1016/j.drugalcdep.2010.12.008. Epub 2011 Feb 2. PMID 21288660
- [Background] Zemore SE, Kaskutas LA. Development and validation of the Alcoholics Anonymous Intention Measure (AAIM). Drug Alcohol Depend. 2009 Oct 1;104(3):204-11. doi: 10.1016/j.drugalcdep.2009.04.019. Epub 2009 Jul 5. PMID 19581057